CLINICAL TRIAL: NCT06783712
Title: Comparative Study Between Ultrasound-Guided IPACK Block (Interspace Between the Popliteal Artery and the Posterior Capsule of the Knee) with Adductor Canal Block Versus Adductor Canal Block Alone for Postoperative Pain Management in Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS47/2024
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-02

CONDITIONS: The Time Interval Between Injection of the Block and the First Rescue Analgesia Dose Given. Postoperative Pain Assessment Using NRS Score for Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I: Adductor canal block alone (Active Comparator)
  Interventions: Procedure: Adductor canal block
- Group II: IPACK block with Adductor canal block (Active Comparator)
  Interventions: Procedure: Adductor Canal Block (ACB) + iPACK Block

INTERVENTIONS:
Procedure: Adductor canal block — Group I: Patients will receive the ultrasound-guided Adductor canal block (ACB) by the supervisors of the research performed just after skin closure. ACB will be performed under complete aseptic conditions. Using a high frequency (6-15MHz) linear probe of an ultrasound machine (Sonosite turbo M, Bothell, Washington, USA) covered with a sterile sheath and 100 mm needle SonoPlex (B-Braun Medical Inc., Bethlehem, PA, USA). ACB block will be performed while the patient is in a supine position at the point midway between the anterior superior iliac spine and the upper pole of the patella. The adductor canal will be located as a hyperechoic structure beneath the sartorius muscle, 100 mm needle SonoPlex will be advanced with the guidance of ultrasound in an in-plane technique and 20 ml bupivacaine (Marcaine) 0.25% will be injected.
  Arms: Group I: Adductor canal block alone
Procedure: Adductor Canal Block (ACB) + iPACK Block — Group II: The patients will receive ACB by the supervisors of the research just after skin closure as previously described in group I and then an IPACK block will be performed. IPACK block will be performed under complete aseptic precautions using the ultrasound machine with the high-frequency linear probe covered with a sterile sheath and 100 mm needle SonoPlex. IPACK block will be performed while the patient is in a supine position with slight knee flexion, the probe will be applied to the popliteal fossa for identification of the popliteal artery and femur. Then the probe will be distally slided for revealing the two femoral condyles followed by proximal sliding of the probe until the humps of the femoral condyles disappear and the flat metaphysis appear. A needle will be advanced from the lateral aspect and directed across the space between the popliteal artery and femur and once the needle reaches the medial edge of the femur,20 ml bupivacaine 0.25% will be injected incrementally
  Arms: Group II: IPACK block with Adductor canal block

SUMMARY:
The investigators will compare the effectiveness of the interspace between the popliteal artery and posterior capsule of the knee (IPACK) block with adductor canal block versus adductor canal block alone for postoperative analgesia in total knee arthroplasty with consequently improved early ambulation and functional rehabilitation.

DETAILED DESCRIPTION:
A.Preoperative settings:

All patients will undergo preoperative assessment (including full history, clinical examination & routine preoperative laboratory investigations will be done (CBC, INR, PT, PTT, and blood chemistry like liver and kidney functions).

B.Intraoperative settings:

On arrival of the patients to the operative room, electrocardiography, non-invasive blood pressure, and pulse oximetry will be applied. Baseline parameters such as systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), heart rate (HR), and oxygen saturation (SpO2) will be recorded. An intravenous (IV) cannula will be inserted, and 500 cc lactated Ringer will be started intravenously as co-load volume. Premedication of 0.02mg/kg of midazolam IV will be given for sedation. Patients will receive spinal anesthesia by the supervisors of the research using the standard technique in a sitting position under complete aseptic conditions using betadine 10%. Then using 4ml lidocaine 2% for local skin infiltration, then introducing a spinal needle 25G (Mercury TM) till getting cerebrospinal fluid (CSF) flow. After getting the CSF flow 12.5mg of heavy bupivacaine 0.5% (Sunny Pharmaceutical Industries, Egypt) will be injected. Then the patient will lie supine with a slight inclination of the head, and then an assessment of the level of spinal anesthesia will be done using cold touch test.

Group I (Adductor canal group): Patients will receive the ultrasound-guided Adductor canal block (ACB) by the supervisors of the research performed just after skin closure. ACB will be performed under complete aseptic conditions. Using a high frequency (6-15MHz) linear probe of an ultrasound machine (Sonosite turbo M, Bothell, Washington, USA) covered with a sterile sheath and 100 mm needle SonoPlex (B-Braun Medical Inc., Bethlehem, PA, USA). ACB block will be performed while the patient is in a supine position at the point midway between the anterior superior iliac spine and the upper pole of the patella. The adductor canal will be located as a hyperechoic structure beneath the sartorius muscle, 100 mm needle SonoPlex will be advanced with the guidance of ultrasound in an in-plane technique and 20 ml bupivacaine (Marcaine) 0.25% will be injected.

Group II: The patients will receive ACB by the supervisors of the research just after skin closure as previously described in group I and then an IPACK block will be performed. IPACK block will be performed under complete aseptic precautions using the ultrasound machine with the high-frequency linear probe covered with a sterile sheath and 100 mm needle SonoPlex. IPACK block will be performed while the patient is in a supine position with slight knee flexion, the probe will be applied to the popliteal fossa for identification of the popliteal artery and femur. Then the probe will be distally slided for revealing the two femoral condyles followed by proximal sliding of the probe until the humps of the femoral condyles disappear and the flat metaphysis appear. A needle will be advanced from the lateral aspect and directed across the space between the popliteal artery and femur and once the needle reaches the medial edge of the femur, nearly at the level of the popliteal artery, negative aspiration is confirmed and 20 ml bupivacaine 0.25% will be injected incrementally as the needle is withdrawn.

C. postoperative settings Vital data including mean arterial blood pressure, heart rate, and oxygen saturation will be recorded 5 minutes before injection of each block and 5 minutes after injection and postoperatively at intervals of 1, 2, 4, 6, 12, 18 & 24 hours. Postoperative pain will be evaluated by a Numeric Rating Scale for pain (NRS Pain) which is an 11-point scale divided as 0=no pain,1-3(mild pain), 4-7(moderate pain), and 7-10 (severe pain), 0-10 scale will be recorded every hour for the first 6 hours and every 2 hours for the rest of the first 24 hours. The time interval between the time of block injection and the time to the first rescue analgesia required (in case of NRS Pain score ≥4) will be measured. If the NRS Pain score is ≥4, patients will receive pethidine 30 mg IV. The total amount of analgesia that will be received in 24 hours postoperatively will be recorded. Assessing hemodynamic data and side effects such as nausea, vomiting, hypotension or hematoma at site of injection.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* The patient refusal to give written consent.
* Previously known allergy to one of the drugs being used in the study.
* Physical status: ASA grades more than III
* History or evidence of coagulopathy, use of anti-coagulant or anti-platelet therapy.
* Patients with neuromuscular disorders
* Injection site infection.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-09 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The time interval between injection of the block and the first rescue analgesia dose given | 24 hours from block injection

CONTACTS AND LOCATIONS:
Overall Officials: Hager Talal Mohamed, MBBCH, Principal Investigator — Anesthesia Resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF